CLINICAL TRIAL: NCT01780883
Title: Melatonin Dose-effect Relation in Childhood Autism
Acronym: MELADOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Centre Hospitalier Guillaume Régnier, RENNES (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANSM A91245-56
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Childhood Autism
Keywords: melatonin; childhood autism; 6-Sulphatoxymelatonin; autistic disorder; dose-effect relation
MeSH Terms: conditions — Autistic Disorder | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): 5 tablets of placebo once a day, an hour before falling asleep, for 6 weeks.
  Interventions: Drug: Placebo
- 2 mg melatonin (Experimental): 1 tablet of 2mg melatonin and 4 tablets of its placebo once a day, an hour before falling asleep, for 6 weeks.
  Interventions: Drug: melatonin; Drug: Placebo
- 4 mg melatonin (Experimental): 2 tablets of 2mg melatonin and 3 tablets of its placebo once a day, an hour before falling asleep, for 6 weeks.
  Interventions: Drug: melatonin; Drug: Placebo
- 10 mg melatonin (Experimental): 5 tablets of 2mg melatonin once a day, an hour before falling asleep, for 6 weeks.
  Interventions: Drug: melatonin

INTERVENTIONS:
Drug: melatonin
  Other Names: Circadin®
  Arms: 10 mg melatonin; 2 mg melatonin; 4 mg melatonin
Drug: Placebo — Placebo tablets of Circadin®
  Arms: 2 mg melatonin; 4 mg melatonin; Placebo

SUMMARY:
Melatonin is a neurohormone produced from serotonin which promotes sleep. The alterations in central and peripheral serotonin neurobiology and in circadian sleep-wake rhythms observed in autistic disorder suggest abnormalities in melatonin secretion.

Several studies have reported a decrease in melatonin secretion in individuals with autism. Furthermore, nocturnal excretion of 6-Sulphatoxymelatonin (the predominant melatonin metabolite) was significantly negatively correlated with severity of autistic impairments in verbal communication and play. Melatonin could therefore have a therapeutic effect on sleep problems and may play a role in the pathophysiology of autistic disorder.

These data highlight the possible therapeutic interest of an oral administration of melatonin in patients with autistic disorder. Thus, the objective of this clinical trial is to study the relation between the melatonin dose administered and its effect on severity of autistic impairments especially in verbal communication and play.

DETAILED DESCRIPTION:
The hormone melatonin is of interest in autism due to theoretical considerations and reports of altered melatonin production in individuals with autism. Melatonin produced in the pineal gland helps regulate human circadian rhythms including sleep-wake, and is considered as the best measure of circadian rhythms.

Several studies revealed that plasmatic and urinary nocturnal levels of melatonin are significantly lower in individuals with autism (in particular, in prepubertal children) compared to typically developing individuals. In addition, this reduction in nocturnal melatonin was significantly associated with the severity of communication and social interaction impairments, especially in verbal communication and play. Finally, diurnal excretion of melatonin was also found to be decreased in individuals with autistic disorder.

Given these results, administration of melatonin could serve, at least in prepubertal children wih autism, to normalize physiological, developmental and behavioral processes that are influenced by this pineal hormone. A randomized clinical trial is therefore necessary to establish potential therapeutic efficacy of melatonin in autistic disorder and to specify its dose-effect relation. This is the first clinical trial studying the melatonin dose-effect in autism.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal males with autism from 6 to 8 years old, according to the diagnostic criteria of autistic disorder of the WHO (CIM-10), American (DSM-IV-TR) and French (CFTMEA) classifications.
* Verbal language level required for the ADOS (Module 1) (i.e., no verbal language as defined by the ADI-R (autism diagnostic interview-revised) scale).
* Written informed consent of the parents or the legal representative.

Non-inclusion Criteria:

* Treatment by benzodiazepines.
* Treatment by anticonvulsant drugs.
* Treatment by serotoninergic products.
* Hypersensitivity reaction to the active substance or one of the excipients of the product.
* Patient with hereditary galactose intolerance, Lapp lactase deficiency or malabsorption syndrome of glucose and galactose.
* Children who are not able to swallow tablets.

Ages: 6 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Severity of autistic disorder | 6 weeks after the beginning of the treatment.

SECONDARY OUTCOMES:
Severity of autistic impairments | 3 weeks after the beginning of the treatment
  Severity of autistic impairments (global severity of autistic disorder and anxiety) using the ADOS (Autism Diagnostic Observation Scale)
Sleep problems | 3 weeks after the beginning of the treatment
  Sleep problems will be assessed using a parental questionnaire and an actimetry sensor in the child recording
Excretion of the urinary metabolite of melatonin | 3 weeks after the beginning of the treatment
  Diurnal and nocturnal excretion of the urinary metabolite of melatonin (6-Sulphatoxymelatonin)
Severity of autistic impairments | 3 weeks after the beginning of the treatment
  Severity of autistic impairments (global severity of autistic disorder and anxiety) using the ICG scale
Severity of autistic impairments | 6 weeks after the beginning of the treatment
  Severity of autistic impairments (global severity of autistic disorder and anxiety) using the ADOS (Autism Diagnostic Observation Scale)
Sleep problems | 6 weeks after the beginning of the treatment
  Sleep problems will be assessed using a parental questionnaire and an actimetry sensor in the child recording
Excretion of the urinary metabolite of melatonin | 6 weeks after the beginning of the treatment
  Diurnal and nocturnal excretion of the urinary metabolite of melatonin (6-Sulphatoxymelatonin)
Severity of autistic impairments | 6 weeks after the beginning of the treatment
  Severity of autistic impairments (global severity of autistic disorder and anxiety) using the ICG scale

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie TORDJMAN, MD, PhD, Principal Investigator — Centre Hospitalier Guillaume Régnier, RENNES; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (4):
- France (4):
  - Service de Psychiatrie de l'Enfant et de l'Adolescent - Hôpital de la Pitié-Salpêtrière, Paris
  - Centre Hospitalier Spécialisé Henri Laborit, Poitiers
  - Service de Psychothérapie de l'Enfant et de l'Adolescent - Hôpital Robert Debré, Reims
  - Pôle de Psychiatrie de l'Enfant et de l'Adolescent - Centre Hospitalier Guillaume Régnier, Rennes

REFERENCES:
- [Result] Tordjman S, Chokron S, Delorme R, Charrier A, Bellissant E, Jaafari N, Fougerou C. Melatonin: Pharmacology, Functions and Therapeutic Benefits. Curr Neuropharmacol. 2017 Apr;15(3):434-443. doi: 10.2174/1570159X14666161228122115. PMID 28503116